CLINICAL TRIAL: NCT02290587
Title: Study of Social Cognition by Morphological and Functional Imaging in Multiple Sclerosis Patients
Acronym: SOCOG-MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: La Ligue Française Contre la Sclérose en Plaques (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2014/01
Record Dates: First submitted 2014-11-05; First posted 2014-11-14 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Multiple Sclerosis
Keywords: social cognitive; theory of mind; cognitive impairment; functional MRI; brain activation network
MeSH Terms: conditions — Multiple Sclerosis; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient (Experimental): MS diagnosis according to McDonald criteria (Polman et al., 2005). Relapsing-remitting MS (RRMS) according to Lublin et al. (1996);
  Interventions: Other: Brain MRI - Clinical and cognitive evaluation; Device: MRI
- Control (Experimental): healthy subject
  Interventions: Other: Brain MRI - Clinical and cognitive evaluation; Device: MRI

INTERVENTIONS:
Other: Brain MRI - Clinical and cognitive evaluation — Neuropsychological evaluation :
  * Questionnaire for depression and anxiety
  * Evaluation of executive functions
  * Evaluation of attention, information processing speed, verbal memory and working memory
  Theory of mind evaluation
  Clinical Evaluation
  MRI Evaluation :
  * morphological MRI
  * functional MRI with two tasks of theory of mind : eyes test and test of attribution of intention
Device: MRI

SUMMARY:
In recent years, studies have brought knowledge of the difficulties of social cognition in Multiple Sclerosis (MS). The brain tissue alteration at the origin of these difficulties in social cognition mechanisms remain poorly understood. Although recent behavioral studies indicated social disturbances in many of these patients, functional studies investigating specific theory of mind in MS are lacking. The use of new techniques for morphological and functional Magnetic Resonance Imaging (MRI) can identify brain activation networks, mapping the achievement and tissue integrity may be related to disorders of social cognition and cognitive. The investigators propose to study social cognition in MS patients using morphological and functional imaging to determine the mechanisms underlying phenomena such as cerebral compensation and its relationship with cognitive impairment.

ELIGIBILITY:
Inclusion Criteria (patient group):

* Aged 18-59 years
* Right handed
* Fluent French speaker
* MS diagnosis according to McDonald criteria (Polman et al., 2005).
* Relapsing-remitting MS (RRMS) according to Lublin et al. (1996);
* Having signed an informed consent (later than the day of inclusion and before any examination required by research)
* Being affiliated to health insurance

Inclusion Criteria (healthy control):

* Aged 18-59 years
* Right handed
* Fluent French speaker
* Having signed an informed consent (later than the day of inclusion and before any examination required by research)
* Being affiliated to health insurance

Exclusion Criteria (patient group):

* Other progressive neurological disease;
* psychiatric comorbidity including severe depression according to Diagnostic and Statistical Manual-IV (DSM-IV),
* alcohol or other addiction to toxic,
* Expanded Disability Status Scale (EDSS) > 6; disabling visual or motor problems preventing participation to neuropsychological assessments,
* relapse since less than one month,
* change of disease-modifying therapy or psychotropic drug since less than one month,
* Contra-indication to MRI (pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin or body, claustrophobia) or refusing MRI
* Illiteracy, is unable to count or to read
* Pregnant or breastfeeding women
* Being under guardianship

Exclusion Criteria (healthy control):

* History of neurological disease;
* family history of MS;
* psychiatric comorbidity including severe depression according to DSM-IV;
* alcohol or other toxic addiction;
* psychotropic drugs; known cognitive complaint or neuropsychological affection;
* Prior neuropsychological testing with the same tests less than one year
* Contra-indication to MRI (pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin or body, claustrophobia) or refusing MRI
* Illiteracy, is unable to count or to read
* Pregnant or breastfeeding women
* Being under guardianship

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Brain activation networks during MRI | At inclusion (day 0)
  To identify brain activation networks during the two paradigms of theory of mind and executive function in RRMS patients taking into account cognitive impairment.

SECONDARY OUTCOMES:
Reduction of volume of deep brain structures and reduction of cortical thickness | At inclusion (day 0)
  Correlation between social cognitive z scores and atrophy measures (reduction of volume of deep brain structures and reduction of cortical thickness).
White matter skeleton on Fractional Anisotropy (FA) maps established by voxel-based. | At inclusion (day 0)
  Comparison of white matter skeleton on Fractional Anisotropy (FA) maps established by voxel-based between RRMS patients and Healthy Control (HC) patients and in RRMS group taking into account cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Brochet, Prof., Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France